CLINICAL TRIAL: NCT02952573
Title: A Phase II Open Label, Multicenter, Trial of JNJ-42756493 In Combination With Dexamethasone For The Treatment Of FGFR3 Wild-type Or Mutation Positive Relapsed and/or Refractory Multiple Myeloma
Brief Title: Testing JNJ-42756493 In Combination With Dexamethasone in Multiple Myeloma That Came Back After a Period of Improvement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low patient accrual
Sponsor: University Health Network, Toronto (Other)
Collaborators: Multiple Myeloma Research Consortium (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM-MM003
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma; Relapsed/Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — erdafitinib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FGFR3 wild-type (Experimental): JNJ-42756493: For the first cycle, 8 mg orally (by mouth), once each day for 14 days of each 28-day periods called cycles. Then dose of JNJ-42756493 may then be increased to 9 mg taken orally if no significant side effects related to JNJ-42756493 are seen during the first 14 days.
  Dexamethasone: 40 mg, orally, on days 1-4, 9-12, 17-20 for the first two cycles. Starting cycle 3, dexamethasone will be taken on days 1, 8, 15 and 22 (once weekly).
  Patients over the age of 75 will take a reduced dose of dexamethasone of 20 mg on starting cycle 1 on days 1-4, 9-12, 17-20 for the first two cycles. Starting cycle 3, dexamethasone will be taken on days 1, 8, 15 and 22 (once weekly).
  Interventions: Drug: JNJ-42756493; Drug: Dexamethasone
- FGFR3 mutated (Experimental): JNJ-42756493: For the first cycle, 8 mg orally (by mouth), once each day for 14 days of each 28-day periods called cycles. Then dose of JNJ-42756493 may then be increased to 9 mg taken orally if no significant side effects related to JNJ-42756493 are seen during the first 14 days.
  Dexamethasone: 40 mg, orally, on days 1-4, 9-12, 17-20 for the first two cycles. Starting cycle 3, dexamethasone will be taken on days 1, 8, 15 and 22 (once weekly).
  Patients over the age of 75 will take a reduced dose of dexamethasone of 20 mg on starting cycle 1 on days 1-4, 9-12, 17-20 for the first two cycles. Starting cycle 3, dexamethasone will be taken on days 1, 8, 15 and 22 (once weekly).
  Interventions: Drug: JNJ-42756493; Drug: Dexamethasone

INTERVENTIONS:
Drug: JNJ-42756493 — Once daily dosing
  Other Names: Erdafitinib
Drug: Dexamethasone — Cycle 1 and 2: OD dosing on days 1-4, 9-12, and 17-20;Cycle 3: OD dosing on days 1, 8, 15, 22
  Other Names: Apo- Dexamethasone

SUMMARY:
This is a phase 2 study to see how effective investigational drug, JNJ-42756493, is when given in combination with dexamethasone in two groups of patients with multiple myeloma (cancer of the plasma cells, a type of white blood cell present in bone marrow) that has relapsed (has come back after a period of improvement) or refractory (did not respond to standard treatment).

DETAILED DESCRIPTION:
Participants in the study will be assigned to one of two groups: One group of participants will be FGFR3 wild-type (participants whose tumors have no mutations or changes of a gene called FGFR3) and the other group will be FGFR3 mutated (participants whose tumors have mutations of FGFR3).

Participants will receive JNJ-42756493 with dexamethasone for as long as their diseases do not progress (worsen) and they do not experience unacceptable side effects for a maximum of 24 cycles (approximately 22 months).

While on the study drugs, participants will be asked to visit the clinic about 2 times during Cycles 1 and 2 and once during Cycle 3 and subsequent cycles for tests and procedures.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of MM and documentation of at least 1 prior line of therapy including proteasome and immunomodulatory agents.
* Documented lab results confirming FGFR3 expression and mutational status determined by a clinical grade, next generation sequencing platform approved by the Sponsor-Investigator, the results of which must be obtained prior to registration.
* Patients with measurable disease by laboratory studies for determining eligibility must be obtained within 28 days prior to start of study drug):
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status score 0, 1, or 2.
* Negative pregnancy status in women of childbearing potential must be confirmed within 7 days prior to start of study drug. Participants must use medically acceptable methods of birth control before the study entry, during the study, and until 3 months after taking the last dose of the study drug.
* Patient must sign the informed consent documents indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Life Expectancy of ≥ 3 months.
* Able to take oral medications.
* Acceptable laboratory results must be met within 7 days of first study drug administration.

Exclusion Criteria:

* Patients in whom FGFR3 expression or mutational status cannot be determined.
* Chemotherapy, limited palliative radiotherapy or other anti-myeloma therapy within 14 days prior to the first dose of study drug. In addition, any treatment related toxicity should have recovered < Grade 1 unless deemed to be irreversible.
* Patients who are receiving any other investigational agent.
* Patients with known CNS involvement, plasma cell leukemia or amyloidosis.
* Use of an investigational drug within 21 days or five-half-lives, whichever is shorter but not less than 14 days, preceding the first dose of study drug.
* History of allogeneic stem cell transplant.
* Autologous, peripheral stem cell transplant within 12 weeks of the first dose of study drug.
* Prior major surgical procedure or extensive radiation therapy within 4 weeks of the first dose of study treatment.
* Current use of corticosteroids, with the exception of inhaled or topical steroids.
* Previous or concurrent malignancies are allowed if it is clear that the patient is not symptomatic from the other tumor. The subject must not be receiving active therapy for the other tumor and the other tumor must be considered medically stable.
* Has a history of or current uncontrolled cardiovascular disease.
* Patients with evidence of mucosal or internal bleeding and/or platelet transfusion refractory. Patients cannot use growth factors within 7 days of start of study drug, or transfusion of blood or platelets within 7 days of start of study drug.
* Has impaired wound healing capacity defined as skin/decubitus ulcers, chronic leg ulcers, known gastric ulcers, or unhealed incisions.
* Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluations.
* Any other condition that, in the Investigator's opinion, would contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Received prior FGFR inhibitor treatment or if the subject has known allergies, hypersensitivity, or intolerance to JNJ-42756493 or its excipients.
* Pregnant, breast feeding, or planning to become pregnant within 3 months after the last dose of study drug and males who plan to father a child while enrolled in this study or within 5 months after the last dose of study drug.
* Known HIV or active hepatitis B or C viral infection.
* History of cerebrovascular accident (CVA) within 6 months prior to registration.
* Gastrointestinal abnormalities, including bowel obstruction, inability to take oral medication, requirement for intravenous (IV) alimentation, active peptic ulcer or prior surgical procedures or bowel resection affecting absorption.
* Peripheral neuropathy ≥ Grade 2.
* Has persistent phosphate level >ULN during screening (within 14 days of treatment and prior to Cycle 1 Day 1) despite medical management.
* Any corneal or retinal abnormality likely to increase the risk of eye toxicity.
* Patients that require the following prohibited therapy:

  1. Medicines known to have a risk of causing QTc prolongation and Torsades de Pointes
  2. Medications known to increase serum levels of phosphate and calcium
  3. Medications or substances known to be strong inhibitors or strong inducers of CYP3A4 or CYP2C9 before the recommended 5 half-life washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 5 years
Minimal response rate | 5 years
Stable disease rate | 5 years

SECONDARY OUTCOMES:
Incidence of toxicities | 5 years
Progression free survival rate | 5 years
Duration of response rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Trudel, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Croucher DC, Devasia AJ, Abelman DD, Mahdipour-Shirayeh A, Li Z, Erdmann N, Tiedemann R, Pugh TJ, Trudel S. Single-cell profiling of multiple myeloma reveals molecular response to FGFR3 inhibitor despite clinical progression. Cold Spring Harb Mol Case Stud. 2023 May 9;9(2):a006249. doi: 10.1101/mcs.a006249. Print 2023 Apr. PMID 36639200